CLINICAL TRIAL: NCT06891443
Title: A Double-Masked, Randomized, Placebo-Controlled, Paired-Eye Study to Evaluate the Efficacy, Safety and Tolerability of Sepofarsen in Subjects With Leber Congenital Amaurosis (LCA) Due to the c.2991+1655A>G (p.Cys998X) Mutation in the CEP290 Gene
Brief Title: Study to Evaluate Sepofarsen in Subjects With Leber Congenital Amaurosis (LCA) Type 10 (HYPERION)
Acronym: HYPERION
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratoires Thea (Industry)
Collaborators: Sepul Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SB-110-007; 2024-518378-14-00 (EU CTIS Number)
Record Dates: First submitted 2025-02-03; First posted 2025-03-24 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-09

CONDITIONS: Leber Congenital Amaurosis 10; Blindness; Leber Congenital Amaurosis; Sensation Disorders; Vision Disorder; Neurological Manifestations; Eye Diseases, Hereditary; Eye Diseases; Eye Disorders Congenital; Retinal Disease
Keywords: LCA10; p.Cys998X; Antisense oligonucleotides; RNA therapy; QR-110; sepofarsen; CEP290; Leber's Congenital Amaurosis; c.2991+1655A>G
MeSH Terms: conditions — Leber Congenital Amaurosis 10; Blindness; Leber Congenital Amaurosis; Sensation Disorders; Vision Disorders; Neurologic Manifestations; Eye Diseases, Hereditary; Eye Diseases; Eye Abnormalities; Retinal Diseases; Meckel Syndrome, Type 4; Optic Atrophy, Hereditary, Leber

STUDY DESIGN:
Intervention Model Description: Paired-eye design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Sepofarsen - Treatment Eye - up to Month 12 (Active Comparator): Subjects to receive Sepofarsen in one eye (160µg first then 40µg) and Placebo in the fellow eye at baseline and at month 6.
  Interventions: Drug: sepofarsen
- Placebo - Fellow Eye - up to Month 12 (Placebo Comparator): Subjects to receive Sepofarsen in one eye (160µg first then 40µg) and Placebo in the fellow eye at baseline and at month 6.
  Interventions: Other: Placebo IVT
- Continued - Treatment Eye - up to Month 24 (Active Comparator): Subjects to receive Sepofarsen (40µg) in one eye and Placebo in the fellow eye at Month 12 and Month 18.
  Interventions: Drug: sepofarsen
- Continued - Fellow Eye - up to Month 24 (Placebo Comparator): Subjects to receive Sepofarsen (40µg) in one eye and Placebo in the fellow eye at Month 12 and Month 18.
  Interventions: Other: Placebo IVT
- Mixed - Treatment Eye - up to Month 24 (Active Comparator): Subjects to receive Sepofarsen (40µg) in one eye and Sepofarsen in the fellow eye (160µg first then 40µg) at Month 12 and at Month 18.
  Interventions: Drug: sepofarsen
- Mixed - Fellow Eye - Month 12 to Month 24 (Active Comparator): Subjects to receive Sepofarsen (40µg) in one eye and Sepofarsen in the fellow eye (160µg first then 40µg) at Month 12 and at Month 18.
  Interventions: Drug: sepofarsen
- Mixed - Fellow Eye - up to Month 12 (Placebo Comparator): Subjects to receive Sepofarsen (40µg) in one eye and Sepofarsen in the fellow eye (160µg first then 40µg) at Month 12 and at Month 18
  Note: up to Month 12 these subjects receive placebo in the Fellow Eye, as all subjects do.
  Interventions: Other: Placebo IVT

INTERVENTIONS:
Drug: sepofarsen — RNA antisense oligonucleotide for intravitreal injection
  Other Names: QR-110
  Arms: Continued - Treatment Eye - up to Month 24; Mixed - Fellow Eye - Month 12 to Month 24; Mixed - Treatment Eye - up to Month 24; Sepofarsen - Treatment Eye - up to Month 12
Other: Placebo IVT — Placebo with identical appearance to sepofarsen
  Arms: Continued - Fellow Eye - up to Month 24; Mixed - Fellow Eye - up to Month 12; Placebo - Fellow Eye - up to Month 12

SUMMARY:
The purpose of this double-masked, randomized, placebo-controlled, paired-eye study is to evaluate the efficacy, safety and tolerability of Sepofarsen in subjects with Leber Congenital Amaurosis (LCA) due to the c.2991+1655A>G (p.Cys998X) mutation in the CEP290.

DETAILED DESCRIPTION:
This is a double-masked, randomized, placebo-controlled, paired-eye study in which one eye of each subject will serve as a control.

At the start of the study the two eyes of each subject will be randomized such that one eye receives sepofarsen and the other eye receives placebo for the first year. In the second year, for all subjects, the eye that was randomized to receive sepofarsen will continue to receive sepofarsen. For the eye that was randomized to placebo in the first year, treatment in the second year will be allocated, as follows: 50% of the eyes will continue to receive placebo, and 50% of the eyes will receive sepofarsen.

Sepofarsen and placebo will be administered via intravitreal injection every 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed clinical diagnosis of LCA10 and a molecular diagnosis of homozygosity or compound heterozygosity for the c.2991+1655A>G mutation in CEP290.
2. Adults: >=18 years / Minors: 6 to <18 years.
3. BCVA (FrACT) equal to or worse than logMAR +0.4 (approximate Snellen equivalent 20/50) to +2.9 logMAR based on quantifiable, reliable FrACT. LP subjects with documented evidence of prior better vision eligible.
4. Symmetrical disease between the two eyes as defined by a BCVA (FrACT) within 0.2 logMAR at baseline.
5. Detectable ONL in the macular area as determined by the CRC at Screening.

Exclusion Criteria:

1. Mutations in genes other than the CEP290 gene associated with other IRD diseases or syndromes.
2. Presence of any ocular pathology in either eye that may make comparison of the eyes not feasible.
3. Presence of unstable concurrent CME, or subject started on (or changed dose of) topical or systemic carbonic anhydrase inhibitor treatment in the 3 months prior to enrollment. CME is allowed if stable for 3 months (with or without treatment).
4. Presence of any clinically significant lens opacities/cataracts based on the AREDS lens grading scale.
5. Any prior receipt of genetic or stem-cell therapy for ocular or non-ocular disease.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Best-Corrected Visual Acuity (BCVA) | 12 Months
  Change from baseline in BCVA based on the Freiburg Acuity and Contrast Test (FrACT) between Treatment Eyes (TEs) and Placebo Control Eyes (PCEs)

SECONDARY OUTCOMES:
Change from baseline in Low Luminance Visual Acuity (LLVA) based on FrACT between Treatment Eyes (TEs) and Placebo Control Eyes (PCEs) | Month 12
Change from baseline in retinal sensitivity as measured by dark-adapted Full-Field Stimulus Test (FST) between Treatment Eyes (TEs) and Placebo Control Eyes (PCEs) | Month 12
Eye-specific Patient Global Impression of Change (PGI-C) between Treatment Eyes (TEs) and Placebo Control Eyes (PCEs) | Month 12
  PGI-C (PATIENT GLOBAL IMPRESSION OF CHANGE ) assesses a patient's perception of overall change in their vision in the respective eye over time. The minimum score (best outcome) is 1 ("Very Much Better") and the maximum score (worst outcome) is 7 ("Very Much Worse"). Higher scores indicate a worse health outcome (greater worsening).
Change from baseline in Contrast Sensitivity (CS) between Treatment Eyes (TEs) and Placebo Control Eyes (PCEs) based on qCSF | Month 12
Change from baseline in retinal sensitivity as measured by light-adapted Full-Field Stimulus Test (FST) between Treatment Eyes (TEs) and Placebo Control Eyes (PCEs) | Month 12
Response in BCVA (FrACT), defined as an improvement of at least 0.2 logMAR from baseline at 12 months and compared between Treatment Eyes (TEs) and Placebo Control Eyes (PCEs), evaluated by the percentage of eyes that achieve this improvement. | Month 12
Response in BCVA (FrACT), defined as an improvement of at least 0.3 logMAR from baseline at 12 months and compared between Treatment Eyes (TEs) and Placebo Control Eyes (PCEs), evaluated by the percentage of eyes that achieve this improvement. | Month 12
Response in Low Luminance Visual Acuity (LLVA) defined as clinically relevant improvement between Treatment Eyes (TEs) and Placebo Control Eyes (PCEs) at 12 months, evaluated by the percentage of eyes that achieve this improvement. | Month 12
Response in Full-Field Stimulus Test (FST) defined as clinically relevant improvement between Treatment Eyes (TEs) and Placebo Control Eyes (PCEs) at 12 months, evaluated by the percentage of eyes that achieve this improvement. | Month 12
Response in Patient Global Impression of Change (PGI-C) defined as clinically relevant improvement between Treatment Eyes (TEs) and Placebo Control Eyes (PCEs) at 12 months, evaluated by the percentage of eyes that achieve this improvement. | Month 12
Response in Contrast Sensitivity (CS) defined as clinically relevant improvement between Treatment Eyes (TEs) and Placebo Control Eyes (PCEs) at 12 months, evaluated by the percentage of eyes that achieve this improvement. | Month 12
Change from baseline in the Michigan Retinal Degeneration Questionnaire (MRDQ) score for subjects ≥ 13 years of age | Month 12
Change from baseline in the Michigan Vision-Related Anxiety Questionnaire (MVAQ) score for subjects ≥ 13 years of age | Month 12
Change from baseline in the Pediatric Eye Questionnaire (PedEyeQ) score for subjects < 13 years of age | Month 12
Change from baseline in eye-specific Patient Global Impression of Severity (PGI-S) between Treatment Eyes (TEs) and Placebo Control Eyes (PCEs) | Month 12
  PGI-S (PATIENT GLOBAL IMPRESSION OF SEVERITY ) assesses a patient's perception of severity of their eye condition in the respective eye over the past week. The minimum score (best outcome) is 1 ("None") and the maximum score (worst outcome) is 5 ("Very Severe"). Higher scores indicate a worse health outcome (greater severity).
Change from baseline in Best-Corrected Visual Acuity (BCVA) based on the ETDRS or the BRVT between Treatment Eyes (TEs) and Placebo Control Eyes (PCEs) | Month 12
Change from baseline in Low Luminance Visual Acuity (LLVA) based on the ETDRS or the BRVT between Treatment Eyes (TEs) and Placebo Control Eyes (PCEs) | Month 12

CONTACTS AND LOCATIONS:
Locations (13):
- United States (5):
  - UCSF Wayne and Gladys Valley Center for Vision, San Francisco, California
  - University of Miami - Bascom Palmer Eye Institute, Miami, Florida
  - University of Iowa, Iowa City, Iowa
  - University of Minnesota Medical School, Minneapolis, Minnesota
  - University of Pennsylvania - Center for Advanced Retinal & Ocular Therapeutics, Philadelphia, Pennsylvania
- Universitair Ziekenhuis Gent (UZ), Ghent, Belgium
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - The Hospital for Sick Children - SickKids, Toronto, Ontario
- Centre de maladies rares CHNO des Quinze Vingt, Paris, France
- Germany (2):
  - Justus-Liebig Universität - Department of Ophthalmology, Giessen
  - University of Tuebingen - Inst. for Ophthalmic Research, Tübingen
- Radboud Universitair Medisch Centrum, Nijmegen, Netherlands
- Moorfields Eye Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No